CLINICAL TRIAL: NCT06133127
Title: Is There an Association Between Quadriceps Strength and Different Markers of Fragility in Patients With Cirrhosis?
Acronym: FRACIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2023 ABERGEL; 2023-A01460-45 (Other: ANSM)
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Cirrhosis
Keywords: Frailty markers; Quadriceps strength
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cirrhosis (45) (Other): Same assessments for all patients (cirrhosis)
  Interventions: Other: Frailty assessment
- Healthy volunteers (15 subjects) (Other): Same assessments for all healthy volunteers
  Interventions: Other: Frailty assessments

INTERVENTIONS:
Other: Frailty assessment — Assessments for all patients : isometric quadriceps strength, malnutrition by RFH-NPT and MNA questionnaires, body composition by circumference and triceps skinfold, frailty by LFI and SPPB, muscle cramps by Cramp questionnaire.
  Arms: Patients with cirrhosis (45)
Other: Frailty assessments — Assessments for all healthy volunteers: isometric quadriceps strength, body composition by circumference and triceps skinfold, frailty by LFI and SPPB.
  Arms: Healthy volunteers (15 subjects)

SUMMARY:
Physical frailty and malnutrition are important factors in morbidity and mortality in patients with cirrhosis. No study has assessed the validity of Liver Frailty Index (LFI) against reference measures such as maximal lower limb strength.

Main objective: To assess the association between LFI score and isometric maximal lower limb strength (quadriceps) in patients with cirrhosis.

DETAILED DESCRIPTION:
Secondary objective: compare the different strength parameters of patients with cirrhosis (strength endurance, rate of strength development) with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

SUBJECT :

* with a diagnosis of liver cirrhosis (regardless of cirrhosis stage and etiology)
* under the care of a physician practising in the University Hospital Estaing in Clermont-Ferrand
* affiliated to the french social security system

Exclusion Criteria:

SUBJECT:

* with hepatocellular carcinoma
* with HIV infection
* with hepatic encephalopathy grade ≥ 2
* with cognitive dysfunction
* with contraindication for physical activity
* with knee pain/knee disorders
* pregnant or breastfeeding
* under protective supervision (guardianship, curatorship, protection of the court)

Inclusion Criteria for healthy volonteers:

* male subjects aged 52 to 62
* female subjects aged 42 to 60
* BMI between 20 and 30 kg/m2
* no musculoskeletal problems limiting physical activity
* level of physical activity < 3 hours per week
* affiliated to the french social security system

Exclusion Criteria for healthy volonteers:

* medical or surgical history deemed incompatible with the trial by the investigator
* simultaneous participation in a trial involving a drug or medical device, or period of exclusion from such a trial
* participants protected by law (under guardianship, conservatorship, or protection of the court)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Isometric quadriceps strength | once, at inclusion
  Isometric quadriceps strength (N.m) will be assessed 3 times with 30 second rest between each try. The dominant leg of each participant will be assessed, a standardised warm-up will be conducted to have effective results.

SECONDARY OUTCOMES:
Malnutrition: Royal Free Hospital-Nutritional Prioritizing Tool (RFH-NPT) | once, at inclusion
Malnutrition: Mini Nutritional Assessment (MNA)) | once, at inclusion
Body composition by circumference and triceps skinfold | once, at inclusion
Frailty by LFI | once, at inclusion
Frailty by Short Physical Performance Battery (SPPB) | once, at inclusion
Muscle cramps by Cramp questionnaire | once, at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Armando ABERGEL, Principal Investigator — aabergel@chu-clermontferrand.fr
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided